CLINICAL TRIAL: NCT05318521
Title: A Randomized, Double-Blind, Parallel-Arm Study Comparing the Efficacy of Investigational Product "Ibuprofen Modified-Release Tablets 800 mg" and Placebo in Patients With Chronic Pain Related to Osteoarthritis of the Knee
Brief Title: RCT, Blinded, 2-Arm Efficacy Study of IP and Placebo in Patients With Chronic Pain Related to Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OVEIBUA20201225
Record Dates: First submitted 2021-12-20; First posted 2022-04-08 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-12

CONDITIONS: Degenerative Arthritis
Keywords: Ibuprofen Modified-Release Tablets; chronic pain related to osteoarthritis of the knee; general pain; fast onset and longer effectiveness
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Approximately 500 evaluable patients will be enrolled. The randomized, IP-treated subject with baseline value for primary analysis will be considered evaluable. Considering an estimated randomization failure rate of 10%, approximately 556 eligible patients will be recruited. Eligible patients will be randomly assigned to receive IBUMR or placebo at a fixed ratio of 1:1. The treatment regimen will be dosing twice a day (BID) for a total of 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen Modified-Release Tablets 800 mg (IBUMR) (Active Comparator): Ibuprofen Modified-Release Tablets 800 mg (IBUMR), twice daily with 12h interval, for 12-week treatment period.
  Interventions: Drug: Ibuprofen modified release tablet 800 mg
- placebo (Placebo Comparator): placebo 800mg, twice daily with 12h interval, for 12-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — The 800mg ibuprofen sustained-release tablet is the same as the next generation of ibuprofen sustained-release tablets developed by foreign pharmaceutical companies, but does not contain a placebo that the active ingredient of ibuprofen
  Other Names: IBUMR
  Arms: placebo
Drug: Ibuprofen modified release tablet 800 mg — Medication: ibuprofen modified sustained release tablets 800 mg Ibuprofen sustained Release Tablet 800mg is a new generation of ibuprofen developed by overseas pharmaceutical companies. It works fast and lasts for up to 12 hours. The dosing regimen was twice daily, 12 hours apart. Ibuprofen :2-[4-(2-methylpropyl) phenyl] propionic acid, nonselective nonsteroidal anti-inflammatory drug (NSAID).
  Other Names: IBUMR
  Arms: Ibuprofen Modified-Release Tablets 800 mg (IBUMR)

SUMMARY:
It is a Phase III efficacy study as the title 'A randomized, double-blind, parallel-arm study comparing the efficacy of investigational product "Ibuprofen Modified-Release Tablets 800 mg" and placebo in patients with chronic pain related to osteoarthritis of the knee.' The primary objective is to determine the analgesic efficacy of orally administered IBUMR in patients with osteoarthritis (OA) of the knee.

The Secondary objectives are to compare the treatment effect on patient pain, function and stiffness between IBUMR- and placebo-treated patients as measured by the Western Ontario and McMaster Osteoarthritis Index (WOMAC), to compare the treatment effect on Patient Global Assessment on Disease Activity between IBUMR- and placebo-treated patients, to compare the treatment effect on Investigator's Global Assessment on Disease Activity between IBUMR- and placebo-treated patients, to compare the use of analgesic rescue medicine between IBUMR- and placebo-treated patients, to determine the safety profile of IBUMR.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded, placebo-controlled, parallel group-study. The duration will be approximately 127 days (4 weeks screening; 12 weeks treatment; 2 weeks follow-up. Currently, Approximately 9 sites in Taiwan and 6 sites in the United States have been selected. Approximately 500 evaluable patients will be enrolled and randomly assigned to receive IBUMR or placebo at a fixed ratio of 1:1. The treatment regimen will be dosing twice a day (BID) for a total of 12 weeks.. The randomized, IP-treated subject with baseline value for primary analysis will be considered evaluable. Considering an estimated randomization failure rate of 10%, approximately 556 eligible patients will be recruited.

For Primary Endpoint, WOMAC Pain will be measured using visual analogue scale (VAS) ranging from 0 mm (no pain) to 100 mm (extreme pain) at baseline week (Day -6 to Day 1) and at Day 8, 15, 22, 29, 43, 57 and Week 12 (Day 79 to Day 85).

For secondary endpoint, WOMAC Physical function will be measured using VAS ranging from 0 mm (no difficulty) to 100 mm (extreme difficulty) at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85. WOMAC stiffness will be measured using VAS ranging from 0 mm (no stiffness) to 100 mm (maximum stiffness) at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85. WOMAC Total Index will be calculated at baseline (Day 1) and Day 8, 15, 22, 29, 43, 57 and 85 as sum of scores of all 24 WOMAC questions.

For other secondary endpoints, Patients will perform a PGADS via a 0-100 mm VAS, ranging from 0 mm (best ever) to 100 mm (worst ever) with respect to "Considering all the ways your arthritis conditionhas affected you, how do you feel your arthritis is today? " PGADS will be calculated periodically, at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85. The degree of the patient's disease status, based on the Investigator's judgment, in terms of pain intensity, joint swelling and tenderness, functional capacity and ability to flex the knee will be assessed by an established IGADS (0-4 point Likert scale), ranging from 0 (very well) to 4 (very poor). IGADS scores will be calculated periodically, at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85.

Safety will also be monitored and evaluated by changes occurring at the baseline and during treatment periods.

Subjects may withdraw from this study due to reasons. A withdrawal occurs when an enrolled patient ceases to participate in the study, regardless of the circumstances, prior to completion of the protocol. The investigators should try their best to complete the evaluation items for the final evaluation visit upon a patient's withdrawal. The reason for a patient withdrawn from the study will be recorded in the case report form (CRF) and in the patient's medical record.

The sample size of this study was based on results from a previous study (Puopolo et al., 2007(2)) which suggested that the least-square mean (95% CI) change in WOMAC pain scores (WOMAC-PS) from baseline is -24.10 (-27.20, -20.99) for treatment group (2400 mg/day; 800 mg TID) and -16.47 (-20.55, -12.40) for placebo group, respectively.

Considering the regimen of our study product (1600 mg; 800 mg BID) and the primary estimand which imputes efficacy data with baseline values for subjects with intercurrent events, we adjusted the treatment effect to -6.005 which is conditional under a 20% reduction in the treatment effect from the study by Puopolo et al. in 2007 (i.e., -7.63 = -24.10 - (-16.47)) and the effect of data imputation, which the proportions of missing data are assumed to be 15% in treatment group and 20% in control group.

A sample size of 250 in each group will have ≥ 85% power to detect a difference in means of -6.005 between treatment and control groups, assuming that the standard deviation for treatment group (t) is 22.879 and the standard deviation for placebo group (p) is 21.463, using a two group Satterthwaite t-test with a 0.050 two-sided significance level.

Analyses on efficacy endpoints will utilize mITT population. A sensitivity analysis using PP population to analyze efficacy endpoints will be conducted if more than 20% of patients are excluded from PP population. Safety evaluation will be performed on mITT population. The conclusion of efficacy (i.e., primary endpoint analysis) of the study will be made according to the results of mITT analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age at the screening visit.
2. Patients diagnosed with symptomatic OA of the knee based on the American College of Rheumatology (ACR) clinical criteria and have an American Rheumatology Association (ARA) functional class rating of I, II, or III (1), for ≥ 3 months prior to date of screening; with recent (≤ 6 months) radiographic evidence of tibiofemoral OA: ≥ Grade 2 on the Kellgren & Lawrence scale. (In cases where both knees are affected, the most painful knee joint is selected as the target knee for study evaluation).
3. Patients had been prescribed NSAIDs or acetaminophen to treat their OA-related pain for at least 3 months prior to the screening visit.
4. Following discontinuation of analgesic medication (a washout period of at least 5 times the half-life (prior to Day -7), plus a subsequent additional 7 days prior to Baseline visit (Day -7 to Day-1), patients must have a reported pain score of at least 40 mm for WOMAC Pain intensity question: 'walking on a flat surface' at Baseline Visit.
5. Subjects are willing to comply with protocol-stated requirements, instructions and restrictions, followed by understanding and signing the written informed consent form or legal representative if he/she is under the statutory age of consent as per the local authority.

Exclusion Criteria:

1. Patients with a history of gastroduodenal perforations and/or obstructions; gastric and/or duodenal surgery; recent (≤ 6 months) active gastrointestinal (GI) ulceration; inflammatory bowel disease; GI bleeding in the past year.
2. Patients with a history of congestive heart failure, coronary artery disease, renal artery stenosis or recent (within 1 year) myocardial infarction, angina, stroke, or transient ischemic attack and/or with uncontrolled hypertension.
3. Patients with moderate to severe hepatic impairment (alanine aminotransferase [ALT] or aspartate transaminase [AST] concentrations > 2.5 times the upper limit of normal).
4. Patients with a medical condition (e.g., a cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine [adrenal hyperplasia], immunologic, dermatologic, neurologic, oncologic, or psychiatric) or a significant laboratory abnormality that, in the Investigator's opinion, would jeopardize the safety of the patient or is likely to confound the study measurements.
5. Patients receiving ongoing opioid therapy for their OA-related pain; or requiring ongoing use of analgesic therapy for other indications, anticoagulants, psychotherapeutic agents, aspirin at daily doses greater than 325 mg, statin-class hypolipidemic agents at doses that have not been stabilized, or other treatments known to interfere with pain perception. (Note: 'stabilized' is defined as being used for at least 3 months).
6. Patients who have received intra-articular injection of corticosteroids, hyaluronic acid or platelet-rich plasma in the target knee within 6 months prior to the screening visit (within 1 year for long-acting formulations); or have received opioid medication within 14 days prior to the screening visit.
7. Patients who are unable to be prescribed NSAIDs or are known or suspected to have hypersensitivity to study medication or their excipients.
8. Patients who have participated in investigational drug trials and took any investigational therapy within 90 days or a time of 5 half-lives prior to the study dosing.
9. Patients currently pregnant, lactating, or planning to pregnant during the trial period. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods mentioned below, during dosing and for at least 4 weeks after stopping study treatment.

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
   * Combination of any two of the following listed methods: (a+b or a+c, or b+c):

     1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
     3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
10. Subjects with underlying medical, mental, psychological, or other inappropriate conditions that would impair treatment compliance, or in the opinion of the Investigator would not permit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC visual analogue 3.1 Pain intensity subscale, over 12 weeks of treatment. [Time frame: Baseline week up to Week 12] | at baseline week (Day -6 to Day 1) and at Day 8, 15, 22, 29, 43, 57 and Week 12 (Day 79 to Day 85).
  WOMAC Pain will be measured using visual analogue scale (VAS) ranging from 0 mm (no pain) to 100 mm (extreme pain)

SECONDARY OUTCOMES:
1. Change from baseline in WOMAC Physical function subscale of the knee over 12 weeks of treatment. [Time frame: Baseline up to Week 12] | at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85
  WOMAC Physical function will be measured using VAS ranging from 0 mm (no difficulty) to 100 mm (extreme difficulty)
2. Change from baseline in WOMAC Joint stiffness subscale of the knee over 12 weeks of treatment. [Time frame: Baseline up to Week 12] | at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85
  WOMAC stiffness will be measured using VAS ranging from 0 mm (no stiffness) to 100 mm (maximum stiffness)
3. Change from baseline in WOMAC Total Index over 12 weeks of treatment. [Time frame: Baseline up to Week 12] | at baseline (Day 1) and Day 8, 15, 22, 29, 43, 57 and 85 as sum of scores of all 24 WOMAC questions.
  WOMAC Total Index will be calculated

OTHER OUTCOMES:
The ≥ 30% and ≥ 50% responder rate of percent improvement | from baseline to Week 12
  use the WOMAC Pain intensity subscale
Mean change from baseline | over 12 weeks of treatment. [Time frame: Baseline up to Week 12]
  use Patient Global Assessment of Disease Status (PGADS) .a PGADS via a 0-100 mm VAS, ranging from 0 mm (best ever) to 100 mm (worst ever)
Mean change from baseline in IGADS | at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85.
  The degree of the patient's disease status, based on the Investigator's judgment, in terms of pain intensity, joint swelling and tenderness, functional capacity and ability to flex the knee will be assessed by an established IGADS (0-4 point Likert scale), ranging from 0 (very well) to 4 (very poor). IGADS scores will be calculated periodically, at baseline (Day 1) and at Day 8, 15, 22, 29, 43, 57 and 85.
Mean use of rescue medication (daily average number of tablets) | [Time frame: Baseline up to Week 12]
  record and statistically analyse the mean use of rescue medication (daily average number of tablets) for each arm

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Kane, Principal Investigator — Palm Beach Research Center
Locations (1):
- Palm Beach Research Center, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No